CLINICAL TRIAL: NCT06027996
Title: Absorbable Antibacterial Soft Tissue Support in Breast Reconstruction With Infection Outcomes Assessment (ARIA)
Brief Title: Melodi Matrix™ in Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melodi Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01-2023
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Tissue expander implantation with the Melodi Matrix
  Interventions: Device: Absorbable Antibacterial Matrix
- Control (No Intervention): Tissue expander implantation without a matrix

INTERVENTIONS:
Device: Absorbable Antibacterial Matrix — Soft tissue support coated with antibiotics
  Other Names: Melodi Matrix™
  Arms: Treatment

SUMMARY:
Prospective, multicenter, randomized, controlled trial evaluating the safety and effectiveness of an absorbable antibacterial matrix device in two stage prepectoral alloplastic breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Age 22 or older at the time of enrollment.
* Is scheduled to undergo unilateral or bilateral mastectomy (including prophylactic) with immediate two-stage post-mastectomy alloplastic prepectoral breast reconstruction.
* Is able to and willing to comply with the study requirements and providing informed consent.

Exclusion Criteria:

* Has prior history of neoadjuvant radiotherapy.
* Has had prior history of failed tissue expansion or breast implantation at the intended reconstruction site.
* Has an active abscess or infection requiring antibiotics anywhere in their body within 30 days.
* Has a Body Mass Index (BMI) < 14 or > 40.
* Is pregnant or is nursing; or plans to become pregnant during the course of the study.
* Has any connective tissue/autoimmune disorder or rheumatoid disease.
* Has known allergies to study device materials.
* Is participating in another interventional research study that may interfere with study endpoints.
* Has limited life expectancy or co-morbid conditions, social/psychological problems, or cognitive impairments that precludes participation.
* Has a medical condition or is taking medications that would result in elevated risk and/or affect the validity of the study.
* Intraoperative assessment demonstrates unfavorable conditions (i.e., poor mastectomy skin flap thickness or viability) for immediate, two-stage post-mastectomy alloplastic prepectoral reconstruction in any breast.

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Complications of Breast Reconstruction | 6 months
  Key local complications

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Stanford University, Palo Alto, California
  - University of Michigan Health, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, Staten Island, New York
  - The Ohio State University, Columbus, Ohio
  - UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Monument Health, Rapid City, South Dakota
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No